CLINICAL TRIAL: NCT06574841
Title: Effect of Blood Flow Restriction on Pain Perception, Grip Strength and Nerve Conductivity in Patients With Carpal Tunnel Syndrome: A Randomized Controlled Trial.
Brief Title: Effect of Blood Flow Restriction on Pain Perception, Grip Strength and Nerve Conductivity in CTS Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElMelhat, Effect of BFR on Pain perception,Grip Strength and Nerve conductivity in CTS patients, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Blood Flow Restriction (BFR)
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome, Blood Flow Restriction.
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction Training (Active Comparator): Blood flow restriction resistance exercise (BFR-RE) involves partially restricting arterial blood flow and fully restricting venous blood flow in the active limb during exercise, utilizing loads typically set at 20% to 30% of an individual's maximum repetition (1RM). It will conduct 3-5 sets until concentric failure is achieved, each set will contain 15-30 repetitions. Moreover, rest periods will range from 30 to 60 seconds and 3 sessions per week will be performed.
  Interventions: Other: Blood Flow Restriction training
- Conventional Physical therapy (Experimental): It consists of the application of a neural custom volar orthotic device to be worn at night and during strenuous daytime activities. Moreover,exercises required patients to assume five different finger postures during tendon-gliding activities: Straight, Hook Fist, Duck Position, Straight Fist, and Full Fist. As well as, six different postures during nerve-gliding activites: Wrist positioned neutrally with flexed thumb and fingers, Wrist maintained neutrally with extended thumb and fingers, Extended wrist and fingers with the thumb in a neutral position, Extended wrist, fingers, and thumb, Extended wrist, fingers, and thumb with forearm supination, and Extended wrist, fingers, and thumb with forearm supination, accompanied by gentle stretching of the thumb by the therapist.
  All will be done 10rep x 5 sec hold, 3-5 times daily for 5 weeks.
  Interventions: Other: Blood Flow Restriction training

INTERVENTIONS:
Other: Blood Flow Restriction training — BFR training done 3 sessions per week, each session includes low intensity of 20% to 30% of 1RM, 3 sets of 15 to 30 reps with a 30sec resting period done for 6 weeks.Moreover, nerve and tendon-gliding exercises consists of 10 reps with a 5-second hold, 3-5 times done daily for 5 weeks.
  Other Names: Nerve and tendon-gliding exercises with a customized volar orthotic device

SUMMARY:
The goal of this clinical trial is to investigate the effect of blood flow restriction (BFR) on pain perception, grip strength and nerve conductivity in patients suffering from carpal tunnel syndrome (CTS). The main question it aims to answer is:

Does performing blood flow restriction training decrease pain, improve grip strength and does not alter nerve conduction velocity in patients with (CTS)? The participants will be divided into two groups to be compared: Patients in the control group will receive the conventional physical therapy program only. In contrast, participants in the experimental group will receive blood flow restriction (BFR) training in addition to a conventional physical therapy program (which includes an orthotic device, tendon, and nerve-gliding exercises).

DETAILED DESCRIPTION:
Blood flow restriction (BFR) entails a training technique that partially limits arterial blood flow and completely restricts venous blood outflow within the active musculature during physical activity (Patterson SD, Hughes L, Warmington S, et al.). This method is thought to have begun in the 1970s through Dr. Yoshiaki Soto's Kaatsu resistance training. By restricting the outflow of blood from the limb, the resulting lack of oxygen creates conditions that stimulate muscle growth through cellular signaling and hormonal changes, resembling the effects of higher-intensity training with increased resistance (Wortman RJ, Brown SM, Savage-Elliott I, Finley ZJ, Mulcahey MK). Emerging studies indicate that Exercise-induced hypoalgesia (EIH) delineates a transient decrease in pain sensitivity subsequent to physical activity (Hughes, L., & Patterson, S. D. (2020)). Moreover, research indicates that individuals diagnosed with carpal tunnel syndrome (CTS) typically exhibit reduced grip strength (Sasaki T, Makino K, Nimura A, et al). Furthermore, acute application of submaximal blood flow restriction (BFR) for approximately ~ 5 minutes does not influence the magnitude or timing of H wave responses (Mendonca, G.V., et al).

Thus, the investigators hypothesized that performing blood flow restriction training will decrease pain, improve grip strength and does not alter the nerve conduction velocity in patients with carpal tunnel syndrome (CTS).

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed by a physician according to the American Academy of Orthopedic Surgeon with carpal tunnel syndrome (CTS).
2. age:30-55 years old.
3. females.
4. positive clinical provocative tests for CTS (Tinel test and Phalen test).
5. subjects with a history of paresthesia, numbness, or pain in the median nerve distribution, night waking, and nocturnal pain.

Exclusion Criteria:

1. subjects who had carpal tunnel release surgery.
2. subjects with cervical disc prolapse.
3. subjects with cervical spondylosis.
4. subjects with thoracic outlet syndrome (TOS).
5. subjects with diabetes.
6. subjects with gestational diabetes.
7. subjects with cardiovascular disorders.
8. subjects with hypertension.
9. pregnant women.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-12-18 (Estimated); Study Completion 2025-01-27 (Estimated)

PRIMARY OUTCOMES:
Electromyography to evaluate median nerve abnormalities specifically within the wrist, assessing their severity, and ruling out other conditions that may imitate carpal tunnel syndrome. | Baseline and after 6 weeks
  EMG activity for motor and sensory nerve conduction:
  1. Electrode used for motor median nerve conduction positioned over the abductor pollicis brevis.
  2. Electrode used for sensory median nerve conduction positioned 2cm distally for the thumb, the index, middle, and ring finger.

SECONDARY OUTCOMES:
Grip Strength | Baseline and after 6 weeks
  The JAMAR Hydraulic Hand Dynamometer, frequently utilized in research investigations, holds a powerful validation and is esteemed as the gold standard against which the efficacy of other devices is measured.
Numerical pain rating scale | Baseline and after 6 weeks
  The numeric rating scale (NRS) is a widely utilized pain screening tool for assessing the severity of pain at a given moment, utilizing a scale from 0 to 10. Zero denotes the absence of pain, while 10 signifies the highest imaginable pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M El Melhat, Phd, Study Director — Cairo University
Locations (1):
- Ahmed ElMelhat [aelmelhat], Cairo, Egypt

REFERENCES:
- [Result] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Result] Wortman RJ, Brown SM, Savage-Elliott I, Finley ZJ, Mulcahey MK. Blood Flow Restriction Training for Athletes: A Systematic Review. Am J Sports Med. 2021 Jun;49(7):1938-1944. doi: 10.1177/0363546520964454. Epub 2020 Nov 16. PMID 33196300
- [Result] Hughes L, Patterson SD. The effect of blood flow restriction exercise on exercise-induced hypoalgesia and endogenous opioid and endocannabinoid mechanisms of pain modulation. J Appl Physiol (1985). 2020 Apr 1;128(4):914-924. doi: 10.1152/japplphysiol.00768.2019. Epub 2020 Feb 27. PMID 32105522
- [Result] Sasaki T, Makino K, Nimura A, Suzuki S, Kuroiwa T, Koyama T, Okawa A, Terada H, Fujita K. Assessment of grip-motion characteristics in carpal tunnel syndrome patients using a novel finger grip dynamometer system. J Orthop Surg Res. 2020 Jul 6;15(1):245. doi: 10.1186/s13018-020-01773-9. PMID 32631378
- [Result] Mendonca GV, Mouro M, Vila-Cha C, Pezarat-Correia P. Nerve conduction during acute blood-flow restriction with and without low-intensity exercise Nerve conduction and blood-flow restriction. Sci Rep. 2020 Apr 30;10(1):7380. doi: 10.1038/s41598-020-64379-5. PMID 32355236